CLINICAL TRIAL: NCT02234245
Title: Economic Evaluation in Cardiology: Remote Monitoring of Pacemakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Antonio Lopez Villegas, PhD student, Universidad de Almeria
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CEIC-AL 53/2012
Record Dates: First submitted 2014-08-28; First posted 2014-09-09 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Disease
Keywords: Follow-Up studies; Biological Pacemakers; Telemedicine; Efficiency
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital monitoring of pacemakers (No Intervention): Patients have to go to the hospital to be monitorized
- Remote monitoring of pacemakers (Experimental): Telemedicine System:
  Patients have not to go to the hospital to be monitorized
  Interventions: Device: Telemedicine System

INTERVENTIONS:
Device: Telemedicine System — Telemedicine System is used in remote monitoring group
  Other Names: Patients are monitorized from hospital
  Arms: Remote monitoring of pacemakers

SUMMARY:
The purpose of this research is to estimate the outcomes in health and cost of the follow-up of patients with pacemakers.

The initial hypothesize of this study is that remote monitoring of pacemaker will show a best relation of outcomes in costs and effectiveness than the conventional follow-up in hospital.

DETAILED DESCRIPTION:
Cardiovascular Diseases are a major cause of global morbidity and mortality, being responsible according to the World Health Organization of the 30% of overall mortality.

Since 2001 that the first pacemaker of remote monitoring was implanted in Europe, more than 300,000 pacemaker have been implanted around the world. Despite this sharp expansion, the scientific evidence on economic evaluations of pacemaker with remote monitoring is very limited, and in our knowledge, studies including informal costs have not been conducted.

In the field of cardiology, telemedicine allows consultations with patients through monitoring systems and remote communication analyzing the ongoing heart rates of people with pacemakers, implantable cardioverter defibrillators, cardiac resynchronization therapy and subcutaneous Holter. The use of remote monitoring may save time and efforts to both healthcare professionals and patients, including their informal caregivers, reducing the number of follow up visits to the hospital and reducing the associated costs with patient follow-up, which will help to improve sustainability of healthcare services.

During the 12 months of study, the patients with implant of pacemakers of both groups will be assessed of the same parameters, in 4 different moments (pre-implant and months 1, 6, 12 and 5 years post-implantation).

The study will estimate: 1) The Clinical features of the patients. 2) The effectiveness through of administration of health-related quality of life, functional capacity questionnaires and 3) Finally, the hospital and informal costs of patients with pacemakers will be estimated by the researches.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age
* Have a pacemaker implanted
* Understand and be able to properly perform self-monitoring at home

Exclusion Criteria:

* Be participating in another study
* Refuse to participate in the study
* Have implanted a different cardiac device to the pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Clinical features | 12 months
  Selected variables from the medical history records:
  * gender
  * age
  * indication for the implantation of the pacemaker.
  * comorbidities
  * pharmacological treatment
  * vital signs
  * pacemaker parameters

SECONDARY OUTCOMES:
Health-Related Quality of Life | 5 years
  EuroQol-5Dimensions (EQ-5D)
Functional capacity | 5 years
  Duke Activity Status Index (DASI).
Direct costs | 5 years
  Direct costs taken into account:
  * pacemakers' costs´(device implanted)
  * hospitalizations' costs
  * consultations' costs (hospital)
  * prescribed medical transport's cost
  * health personnel costs
  * pharmaceutical costs
Indirect cost | 5 years
  Maintenance of the medical consultation (hospital):
  * electricity
  * cleaning
  * furniture
  * Health fungible
  * equipment investment
Informal costs | 5 years
  Costs related to the care and displacements of patients to hospital:
  * displacement costs to hospital
  * Accommodation costs
  * Cost of meals
  * Costs for caregivers
Number of patients with Adverse Events | 5 years
  Number of patients with Adverse Events
  - type of Adverse Events diagnosed
Consultations and Hospitalizations unscheduled | 5 years
  - number of unscheduled visits and hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Poniente, El Ejido, Almeria, Spain

REFERENCES:
- [Derived] Catalan-Matamoros D, Lopez-Villegas A, Leal Costa C, Bautista-Mesa R, Robles-Musso E, Rocamora Perez P, Lopez-Liria R. A non-randomized clinical trial to examine patients' experiences and communication during telemonitoring of pacemakers after five years follow-up. PLoS One. 2021 Dec 23;16(12):e0261158. doi: 10.1371/journal.pone.0261158. eCollection 2021. PMID 34941904
- [Derived] Bautista-Mesa RJ, Lopez-Villegas A, Peiro S, Catalan-Matamoros D, Robles-Musso E, Lopez-Liria R, Leal-Costa C. Long-term cost-utility analysis of remote monitoring of older patients with pacemakers: the PONIENTE study. BMC Geriatr. 2020 Nov 16;20(1):474. doi: 10.1186/s12877-020-01883-3. PMID 33198629
- [Derived] Lopez-Villegas A, Catalan-Matamoros D, Robles-Musso E, Peiro S. Workload, time and costs of the informal cares in patients with tele-monitoring of pacemakers: the PONIENTE study. Clin Res Cardiol. 2016 Apr;105(4):307-13. doi: 10.1007/s00392-015-0921-5. Epub 2015 Sep 30. PMID 26423396
- [Derived] Lopez-Villegas A, Catalan-Matamoros D, Robles-Musso E, Peiro S. [Comparative Effectiveness of Remote Monitoring of People with Cardiac Pacemaker versus Conventional: quality of Life at the 6 Months]. Rev Esp Salud Publica. 2015 Apr;89(2):149-58. doi: 10.4321/S1135-57272015000200004. Spanish. PMID 26121625